CLINICAL TRIAL: NCT00843141
Title: ADHD Symptoms, Executive Functions and Quality of Life Following Three Months of Training.
Brief Title: The Efficacy of Computerized Cognitive Training in Adults With ADHD: Change in ADHD Symptoms, Executive Functions and Quality of Life Following Three Months of Training.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Prof. Omer Bonne, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADHDA-HMO-CTIL
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2009-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Executive functions; Quality of life
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cognitive computerized training (Experimental): cognitive computerized training utilizing executive attention tasks
  Interventions: Behavioral: cognitive computerized training
- simple cognitive computerized training (Active Comparator): simple computerized cognitive program utilising simple reaction time tasks that do not challenge executive attention
  Interventions: Behavioral: simple cognitive computerized training

INTERVENTIONS:
Behavioral: cognitive computerized training — cognitive computerized training utilizing executive attention tasks
  Arms: cognitive computerized training
Behavioral: simple cognitive computerized training — simple computerized cognitive program utilising simple reaction time tasks that do not challenge executive attention
  Arms: simple cognitive computerized training

SUMMARY:
The study group of Adults with ADHD who will receive cognitive (executive attention) computerized training will show significant improvement in ADHD symptomatology,neuropsychological measures,daily functioning and quality of life.

A significant difference will be found between the study group and the control group (adults with ADHD that will receive a simplified cognitive training program that does not challenge their executive functions)on the above measures.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18-60);
* 9 years education;
* Diagnosis of ADHD;
* Executive function deficit in daily life;
* Signed informed consent.

Exclusion Criteria:

* Change in pharmacological treatment and/or received new treatment for ADHD in the last three months;
* Other current serious neurological disorder (e.g. epilepsy, brain injury, neurodegenerative disease), other major current and sever psychiatric disorder (axisI);
* Color blindness.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Executive functioning | after 3 months of cognitive training

SECONDARY OUTCOMES:
ADHD symptomatology and quality of life | after 3 months of cognitive training

CONTACTS AND LOCATIONS:
Overall Officials: Omer Bonne, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel